CLINICAL TRIAL: NCT00926913
Title: Investigating Optical and Neural Causes of Vision Loss
Status: Withdrawn | Type: Observational
Why Stopped: Project has ended
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: C7002-R
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
With the aging of the population, the prevalence of age-related macular degeneration (AMD) eye disease has resulted in a large number of people suffering from central vision loss. In fact, the most prevalent cause of blindness among veterans is AMD. Since the number of elderly veterans is expected to double in the next 10 years, loss of vision due to AMD is also expected to proportionally and considerably escalate. People with impaired vision have difficulty with daily activities, such as, reading, driving, and recognizing faces. The goal of the research project is to provide information on factors that contribute to visual impairment. This knowledge is necessary for the development of innovative approaches that will optimize the benefit of vision rehabilitation techniques, aimed at improving vision, thus allowing our veterans to maintain function and productivity. The findings from the proposed research will benefit our veterans and all aging people.

DETAILED DESCRIPTION:
Vision loss has become a major public health problem due to the growth and aging of the population. Age-related macular degeneration (AMD) is the most common cause of vision loss in people over 50 years of age. In the United States, over 10 million people have AMD and over 1.6 million people age 50 and older have late-stage advanced AMD. It is well established that AMD patients with central vision loss use preferred retinal loci (PRL) which are peripheral retinal areas adjacent to the fovea for performing daily activities, such as reading. However, even in healthy eyes, peripheral vision is limited due to reduced neural sampling density compared to the fovea. Additionally, the function of the peripheral retina can be further reduced in patients, owing to degenerative disease processes. These neural substrate losses are coupled with losses in the quality of the optical image on the retina. Optical imperfections increase with age and off-axis viewing, compared to viewing along the optical axis of the eye. The combination of these factors plays a significant role in reducing visual performance of patients with eccentric fixation. The long term goal of the project is to improve the visual performance of veterans with central vision loss by development of innovative approaches that will optimize the benefit of vision rehabilitation techniques. In the current proposal, optical and neural losses will be assessed in AMD patients with central vision loss using novel techniques. Increased optical losses due to age and viewing off the optical axis of the eye will be established with wavefront analysis technology. Increased neural losses due to retinal dysfunction at PRL will be determined based on measurement of visual acuity with blurred stimuli. Improvement in reading speed will be evaluated, conditional on neural losses at PRL and/or the stability of PRL, after compensating for optical losses with our adaptive optics system. The findings will provide knowledge of PRL function and stability that is beneficial for improving the outcome of available vision rehabilitation methods that train patients to better use their PRLs. Also, customized correction of optical imperfections of the eye for effectively improving visual performance can be developed as an approach for better vision rehabilitation of patients. Optimizing vision rehabilitation of our veterans will allow them to maintain function and productivity.

ELIGIBILITY:
Inclusion Criteria:

Standard inclusion criteria are:

* qualification for entry into the study based on clinical evaluation,
* competence to understand and willingness to sign an informed consent form and participate in the study,
* pupils that dilate to 5 mm or more.

The inclusion criteria for normal subjects will be:

* corrected visual acuities better than 20/30,
* intraocular pressure less than 21 mm Hg,
* no family history of AMD,
* no history of ophthalmic surgery or neurologic disease,
* no history of diabetes, glaucoma, or a history of elevated intraocular pressure.

The recruitment will ensure that approximately 40 subjects will fall into each of the three age groups, 50 to 60 years, 61 to 70 years, and 71 years and older. One eye of each subject will be selected at random to be included in the study.

Exclusion Criteria:

* Ocular opacities that preclude acquiring a clear fundus photograph or refractive errors greater than 4 diopters.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal healthy subjects and patients diagnosed with age-related macular degeneration and central vision loss will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Ocular aberrations | One time only

CONTACTS AND LOCATIONS:
Overall Officials: Mahnaz Shahidi, PhD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States